CLINICAL TRIAL: NCT04289623
Title: Assessing the Impact of myHealth Rewards Program-related Communications on Enrollment: Replication
Status: Completed | Type: Observational
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0218
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Health Promotion; Wellness Program
Keywords: Prospect theory; Social norms; Social proof; Authority

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Standard email: This email mentions the cost-saving benefits of enrollment by participants who met their 2018 goals. It also includes the message that registration can be completed quickly (in less than five minutes). Finally, it also includes reward incentive information, wherein registering by a March deadline provides qualified recipients with the potential to win prizes. This information is contained in all other emails.
  Interventions: Behavioral: Email
- Loss frame email: In addition to the content of the generic email, the subject line and content of the loss frame email recommends that GHP members not "throw away" a precise dollar amount in savings (over $2,000) by not participating and that they can therefore avoid missing out on substantial gains (i.e., savings) by taking action. This email further frames the reward as something recipients will miss out on if they do not sign up.
  This intervention frames the status quo as a state from which recipients, via inaction, are slated to forfeit a sizable and precise monetary amount to which they should otherwise feel entitled (via loss aversion and the endowment effect). People tend to be risk-seeking in the domain of losses; therefore, this intervention is hypothesized to increase enrollment in the hope of achieving zero loss by meeting program goals, as opposed to a sure loss via inaction.
  Interventions: Behavioral: Email; Behavioral: Loss frame
- Testimonial (medical expert) email: In addition to the content of the generic email, the testimonial (medical expert) email includes a testimonial from a doctor, which notes the personal benefits of myHealth Rewards in terms of managing blood pressure, blood sugar, cholesterol, weight, and stress.
  This intervention shows proof of other people successfully enrolling and benefitting from the program. Specifically, it is an endorsement from a presumed authority figure. Recipients may be more likely to enroll for this program if they see a physician - who would be seen as an authority on health and wellness - talking about the medical benefits of the program. It is unclear in the current context and population if a message from an expert or rank-and-file employee would be more effective.
  Interventions: Behavioral: Email; Behavioral: Testimonial (medical expert)
- Testimonial (rank-and-file) email: In addition to the content of the generic email, the testimonial (rank-and-file) email includes a testimonial from a customer care specialist, which notes the personal benefits of myHealth Rewards in terms of managing blood pressure, blood sugar, cholesterol, weight, and stress.
  This intervention shows proof of other people successfully enrolling and benefitting from the program. Specifically, it is an endorsement from a peer (relative to most Geisinger employees). Recipients may be more likely to enroll for this program if they see a rank-and-file employee talking about the program as this person would be more relatable (relative to a doctor). It is unclear in the current context and population if a message from an expert or rank-and-file employee would be more effective.
  Interventions: Behavioral: Email; Behavioral: Testimonial (rank-and-file)
- Social norms (percentage) email: In addition to the content of the generic email, the social norms (percentage) email will include communication about the percentage of benefit-eligible employees who had already registered for myHealth Rewards.
  This message sets up a descriptive norm, showing that a majority of people are doing a certain behavior. When people see a behavior as the norm, they are more likely to follow it. The use of percentages makes it clear that this behavior is indeed being done by most people in the group. It is unclear in the current context and population if a message using percentages or numbers would be more effective.
  Interventions: Behavioral: Email; Behavioral: Social norms (percentage)
- Social norms (number) email: In addition to the content of the generic email, the social norms (number) email will include communication about the number of benefit-eligible employees who had already registered for myHealth Rewards.
  This message sets up a descriptive norm, showing that a large number of people are doing a certain behavior. When people see a behavior as the norm, they are more likely to follow it. While the use of numbers does not indicate that this behavior is being done by a majority, using a large number can be more convincing just in showing sheer quantity.
  Interventions: Behavioral: Email; Behavioral: Social norms (number)

INTERVENTIONS:
Behavioral: Email — Email
Behavioral: Loss frame — Email
  Other Names: Endowment effect
  Groups: Loss frame email
Behavioral: Testimonial (medical expert) — Email
  Other Names: Authority
  Groups: Testimonial (medical expert) email
Behavioral: Testimonial (rank-and-file) — Email
  Other Names: Social proof
  Groups: Testimonial (rank-and-file) email
Behavioral: Social norms (percentage) — Email
  Other Names: Social proof
  Groups: Social norms (percentage) email
Behavioral: Social norms (number) — Email
  Other Names: Social proof
  Groups: Social norms (number) email

SUMMARY:
The purpose of the study is to evaluate, prospectively, the potential impact on myHealth Rewards wellness program enrollment (prior to the 2020 deadline) of sending different messages via email to Geisinger Health Plan (GHP) members who have not yet enrolled. In particular, this study aims to replicate and extend (with greater sample size and statistical power) the findings from a previous study in which email communication using loss framing language achieved significantly higher click-through rates than a more standard communication, whereas actual enrollment rates were not significantly higher.

DETAILED DESCRIPTION:
The myHealth Rewards wellness program managed by GHP rewards those GHP members who carry their insurance through employment at Geisinger with reduced health insurance premiums over the course of the following year, if members register for the program and have their health measures on file by the enrollment deadline and are then able to meet their health goals by the respective due date. In spite of the potential savings to health plan members and the wellness program's potential to motivate engagement in healthy activities (with consequent improvement in health outcomes), about 23% of eligible existing GHP members did not enroll during the primary 2019 enrollment period, even after receiving promotional email communications and reminders.

Previous work examining myHealth Rewards found that email communication using loss framing language achieved significantly higher click-through rates than a more standard communication, whereas actual enrollment rates were not statistically significantly higher.

The current study aims to analyze de-identified Geisinger Health Plan (GHP) member data, comparing enrollment status (and secondarily, click-through rates) within the 2020 enrollment period across email conditions to which GHP members will be randomly assigned. The main part of this study will compare the effects of a standard, generic communication vs. communication with loss framing, using a larger sample size for adequate statistical power to detect the original difference in enrollment rates as significant, should that difference be real and reliable. Additional conditions are added after this main comparison in order to compare more precisely other pairs of communications conceived in the original study.

The generic email condition will consist of a standard email of the kind that would typically be sent by GHP to encourage enrollment, which includes the average amount saved, the ease of registration, and a reward incentive. The loss framing condition will highlight that respondents are forfeiting savings unless they take action and register. The two testimonial conditions will have a testimonial from a doctor (medical expert condition) or a customer care specialist (rank-and-file condition) about how the program helped them. The two social norms conditions will show the percentage (percentage condition) or number (number condition) of fellow Geisinger members who already signed up. Emails will go out in three waves. For each wave, Geisinger employees who have not already registered at that time will be randomized into one of two groups:

Wave 1: generic email vs. loss framing email

Wave 2: testimonial (expert) vs. testimonial (rank-and-file)

Wave 3: social norms (percentage) vs. social norms (number)

It is hypothesized that, on average, the loss frame email will increase enrollment compared with the standard email. The other comparisons are exploratory and do not have a priori hypotheses. Findings will help inform how best to increase enrollment in a wellness program through email communication.

ELIGIBILITY:
Inclusion Criteria:

* Geisinger Health Plan members
* Geisinger Health System employees who have not yet enrolled in myHealth Rewards

Exclusion Criteria:

* Enrollment in myHealth Rewards before the email launch date for each wave
* Do not have an email address on file

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population consists of Geisinger Health System employees who are also Geisinger Health Plan members and are not currently enrolled in myHealth Rewards.
Sampling Method: Probability Sample
Enrollment: 13546 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings. The PI did not examine or analyze any data from this study prior to this registration.
Supporting Information: Study Protocol
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were sent the Wave 1 emails on February 25, 2020.
Groups:
- Loss Frame Email: In addition to the content of the generic email, the subject line and content of the loss frame email recommends that GHP members not "throw away" a precise dollar amount in savings (over $2,000) by not participating and that they can therefore avoid missing out on substantial gains (i.e., savings) by taking action. This email further frames the reward as something recipients will miss out on if they do not sign up.
- Testimonial (Medical Expert) Email: In addition to the content of the generic email, the testimonial (medical expert) email includes a testimonial from a doctor, which notes the personal benefits of myHealth Rewards in terms of managing blood pressure, blood sugar, cholesterol, weight, and stress.
- Testimonial (Rank-and-file) Email: In addition to the content of the generic email, the testimonial (rank-and-file) email includes a testimonial from a customer care specialist, which notes the personal benefits of myHealth Rewards in terms of managing blood pressure, blood sugar, cholesterol, weight, and stress.
- Social Norms (Percentage) Email: In addition to the content of the generic email, the social norms (percentage) email will include communication about the percentage of benefit-eligible employees who had already registered for myHealth Rewards.
- Social Norms (Number) Email: In addition to the content of the generic email, the social norms (number) email will include communication about the number of benefit-eligible employees who had already registered for myHealth Rewards.
Period: Wave 1 Emails
Arm/Group | Standard Email | Loss Frame Email | Testimonial (Medical Expert) Email | Testimonial (Rank-and-file) Email | Social Norms (Percentage) Email | Social Norms (Number) Email
Started | 6782 | 6764 | 0 (Participants who did not respond to the intervention in Wave 1 were randomly assigned to this intervention or the testimonial (rank-and-file) email in Wave 2.) | 0 (Participants who did not respond to the intervention in Wave 1 were randomly assigned to this intervention or the testimonial (medical expert) email in Wave 2.) | 0 (A planned Wave 3 of the study was not conducted due to COVID-19-related changes in the program being offered as part of the intervention.) | 0 (A planned Wave 3 of the study was not conducted due to COVID-19-related changes in the program being offered as part of the intervention.)
Completed | 6514 | 6507 | 0 | 0 | 0 | 0
Not Completed | 268 | 257 | 0 | 0 | 0 | 0
Not completed — Email was not delivered | 268 | 257 | 0 | 0 | 0 | 0
Period: Wave 2 Emails
Arm/Group | Standard Email | Loss Frame Email | Testimonial (Medical Expert) Email | Testimonial (Rank-and-file) Email | Social Norms (Percentage) Email | Social Norms (Number) Email
Started (The participants who were sent the standard email and the loss frame email but did not respond to the intervention were pooled into one group and randomly assigned to either receive the testimonial (medical expert) email or the testimonial (rank-and-file) email.) | 0 (Participants were already sent this intervention or the loss frame email in Wave 1.) | 0 (Participants were already sent this intervention or the standard email in Wave 1.) | 6099 (Participants who did not respond to the intervention in Wave 1 were randomly assigned to these groups in Wave 2.) | 6117 (Participants who did not respond to the intervention in Wave 1 were randomly assigned to these groups in Wave 2.) | 0 (A planned Wave 3 of the study was not conducted due to COVID-19-related changes in the program being offered as part of the intervention.) | 0 (A planned Wave 3 of the study was not conducted due to COVID-19-related changes in the program being offered as part of the intervention.)
Completed | 0 | 0 | 6099 | 6117 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline outcome measure was not applicable, since enrollment and login in response to the email was the outcome. There was no previous email, and participants were selected for not having enrolled in the year of the study period. The participants who were sent the standard email and the loss frame email but did not respond to the intervention were pooled into one group and randomly assigned to either receive the testimonial (medical expert) email or the testimonial (rank-and-file) email.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Email | Loss Frame Email | Testimonial (Medical Expert) Email | Testimonial (Rank-and-file) Email | Social Norms (Percentage) Email | Social Norms (Number) Email | Total
Number analyzed (Participants) | 6782 | 6764 | 0 | 0 | 0 | 0 | 13546
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Data were not collected. | NA — Data were not collected. | 0 | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | NA — Data were not collected. | NA — Data were not collected. | 0 | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — Data were not collected. | NA — Data were not collected. | 0 | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data were not collected. | NA — Data were not collected. | 0 | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data were not collected. | NA — Data were not collected. | 0 | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6782 | 6764 |  |  |  |  | 13546

OUTCOME MEASURES:

1. Primary Outcome: Rate of Enrollment (14 Days)
Description: Enrollment in the myHealth Rewards program (yes/no) within 14 full days of the beginning of the intervention for each of the three waves.
Time Frame: 14 days
Population: A planned Wave 3 of the study was not conducted due to COVID-19-related changes in the program being offered as part of the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Email | Loss Frame Email | Testimonial (Medical Expert) Email | Testimonial (Rank-and-file) Email | Social Norms (Percentage) Email | Social Norms (Number) Email
Number analyzed (Participants) | 6514 | 6507 | 6099 | 6117 | 0 | 0
Participants
  Previously Enrolled | 540 | 622 | 271 | 258 | 0 | 0
  Never Enrolled | 63 | 52 | 33 | 20 | 0 | 0
Statistical Analysis 1: Comparison: Standard Email vs Loss Frame Email; We conducted a logistic regression among the previously enrolled group with the standard email as the reference group; Test type: Superiority; p = .007, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.05 to 1.35]
Statistical Analysis 2: Comparison: Standard Email vs Loss Frame Email; We conducted a logistic regression among the never enrolled group with the standard email as the reference group; Test type: Superiority; p = .287, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.56 to 1.19]
Statistical Analysis 3: Comparison: Testimonial (Medical Expert) Email vs Testimonial (Rank-and-file) Email; We conducted a logistic regression among the previously enrolled group with the rank-and-file email as the reference group; Test type: Superiority; p = .590, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.87 to 1.27]
Statistical Analysis 4: Comparison: Testimonial (Medical Expert) Email vs Testimonial (Rank-and-file) Email; We conducted a logistic regression among the never enrolled group with the rank-and-file email as the reference group; Test type: Superiority; p = .035, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.05 to 3.32]

2. Primary Outcome: Rate of Logging in (14 Days)
Description: Logging into the myHealth Rewards program (yes/no) within 14 full days of the beginning of the intervention for each of the three waves.
Time Frame: 14 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Email | Loss Frame Email | Testimonial (Medical Expert) Email | Testimonial (Rank-and-file) Email | Social Norms (Percentage) Email | Social Norms (Number) Email
Number analyzed (Participants) | 6514 | 6507 | 6099 | 6117 | 0 | 0
Participants
  Previously Enrolled | 253 | 297 | 47 | 59 | 0 | 0
  Never Enrolled | 48 | 45 | 14 | 15 | 0 | 0
Statistical Analysis 1: Comparison: Standard Email vs Loss Frame Email; We conducted a logistic regression among the previously enrolled group with the standard email as the reference group; Test type: Superiority; p = .085, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.98 to 1.37]
Statistical Analysis 2: Comparison: Standard Email vs Loss Frame Email; We conducted a logistic regression among the never enrolled group with the standard email as the reference group; Test type: Superiority; p = .569, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.60 to 1.33]
Statistical Analysis 3: Comparison: Testimonial (Medical Expert) Email vs Testimonial (Rank-and-file) Email; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = .240, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.54 to 1.17]
Statistical Analysis 4: Comparison: Testimonial (Medical Expert) Email vs Testimonial (Rank-and-file) Email; We conducted a logistic regression among the never enrolled group with the rank-and-file email as the reference group; Test type: Superiority; p = .871, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.45 to 1.95]

ADVERSE EVENTS:
Time Frame: No adverse events were evaluated.
Description: We only received aggregate information about email engagement with no individual-level information collected (including those for adverse events).
Arm/Group | Standard Email | Loss Frame Email | Testimonial (Medical Expert) Email | Testimonial (Rank-and-file) Email | Social Norms (Percentage) Email | Social Norms (Number) Email
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
For this study, we only received data about engagement with the email. Individual patients were not identified and demographic information such as age, sex, or gender were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT04289623/Prot_SAP_000.pdf